CLINICAL TRIAL: NCT02808637
Title: Vaccine-Related Pain in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, İLKNUR GÖL, PhD RN, ASSISTANT PROFESSOR, Çankırı Karatekin University
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CANKIRI KARATEKIN UNIVERSITY
Record Dates: First submitted 2016-06-10; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Pain management; vaccination; manual pressure; needle aspiration
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Manual Pressure (Experimental)
  Interventions: Other: Manual Pressure
- Rapid Injection without Aspiration (Experimental)
  Interventions: Other: Rapid Injection without Aspiration
- Manual Pressure + Rapid Injection without Aspiration (Experimental)
  Interventions: Other: Manual Pressure + Rapid Injection without Aspiration
- Control (Experimental)
  Interventions: Other: Control

INTERVENTIONS:
Other: Manual Pressure — First, the infants were seated on their mothers' knees. Next, 10-second manual pressure was applied on the vaccine injection site. Then DTaP/IPV/Hib was administered in accordance with the conventional injection technique.
  Arms: Manual Pressure
Other: Rapid Injection without Aspiration — First, the infants were seated on their mothers' knees. Then DTaP/IPV/Hib was administered by using rapid injection without aspiration technique.
  Arms: Rapid Injection without Aspiration
Other: Manual Pressure + Rapid Injection without Aspiration — First, the infants were seated on their mothers' knees. Next, 10-second manual pressure was applied on the vaccine injection site. Then DTaP/IPV/Hib was administered by using the rapid injection without aspiration technique.
  Arms: Manual Pressure + Rapid Injection without Aspiration
Other: Control — First, the infants were seated on their mothers' knees. Then DTaP/IPV/Hib was administered by using the conventional injection technique.
  Arms: Control

SUMMARY:
This is a randomized double-blind controlled study and was performed to compare effects of rapid injection without aspiration and 10-second manual pressure before injection on pain severity and crying time in 4-6-month-old infants given the vaccine DTaP/IPV/Hib.

The study population included all the infants presenting for DTaP/IPV/Hib to two family health centers between April and August in 2015. The study sample included 128 infants based on confidence interval of 95% and statistical power of 80%. The sample was divided into four groups; i.e. manual pressure, rapid injection without aspiration, manual pressure combined with rapid injection without aspiration and control groups. There were 32 infants in each group. Gender was adjusted in all groups. Stratified and block randomizations were used.

DETAILED DESCRIPTION:
Study design: this is an experimental, double-blind, randomized controlled trial.

Study population and study sample: The study was conducted in two family health centers of Cankiri Public Health Directorate, Turkey, between April and August in 2015. The study population included infants aged 4-6 months and presenting to the family health centers for the second and third doses of DTaP/IPV/Hib. The study sample comprised of 128 infants based on confidence interval of 95% and statistical power of 80%. Analysis made at the end of the study showed a statistical power of 0.83 based on confidence interval of 95%.

Outcome Measures

Pain severity: Video recordings obtained were evaluated by two pain specialists separately by using Neonatal Infant Pain Scale. The specialists were blinded to the groups to eliminate possible mistakes in observations and the possibility of taking sides and to avoid bias. The scores assigned by the specialists were used to determine pain scores before, during and after vaccine injections.

Crying time: Video recordings taken were watched by the same researcher and crying time before, during and after vaccine injections was calculated for each infant.

Physiological Changes (heart rate and oxygen saturation): the probe of pulse oximetry was attached to the foot not injected vaccine to measure oxygen saturation and heart rate before, during and after the injections in each child.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants who were aged 4-6 months, had the percentiles of 3P - 97P, were born at term and were not given any analgesics before immunization and whose mothers gave written informed consent were included.

Exclusion Criteria:

* Infants whose percentiles were below 3P and above 97P and who had acute infectious diseases, underwent topical anesthesia and/or took analgesics were excluded from the study.

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain severity | 6 MONTHS
  Video recordings obtained were evaluated by two pain specialists separately by using NIPS. The specialists were blinded to the groups to eliminate possible mistakes in observations and the possibility of taking sides and to avoid bias. The scores assigned by the specialists were used to determine pain scores before, during and after vaccine injections. Pain severity, were expressed as the average score NIPS. When the opportunity to observe the baby again during the data collection and it was observed that no adverse effects. Therefore study has been completed with the same 128 babies.
Crying time | 6 MONTHS
  Video recordings taken were watched by the same researcher and crying time (sec) before, during and after vaccine injections was calculated for each infant. When the opportunity to observe the baby again during the data collection and it was observed that no adverse effects. Therefore study has been completed with the same 128 babies.
Physiological Changes (heart rate and oxygen saturation) | 6 MONTHS
  the probe of pulse oximetry was attached to the foot not injected vaccine to measure oxygen saturation (%) and heart rate (min) before, during and after the injections in each child. When the opportunity to observe the baby again during the data collection and it was observed that no adverse effects. Therefore study has been completed with the same 128 babies.